CLINICAL TRIAL: NCT04341220
Title: Additive Effect of Transcranial Direct Current Stimulation on Physiotherapeutic Treatment of Children With Balance Deficit: a Randomized, Controlled, Double-blind Clinical Trial
Brief Title: Effects of Transcranial Direct Current Stimulation on Balance of Children With Balance Deficit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17512619.0.0000.0065
Record Dates: First submitted 2020-03-16; First posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-03

CONDITIONS: Postural Balance
Keywords: Transcranial Direct Current Stimulation; Children; Child Development; Motor Control
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tDCS + Exercise (Experimental): Anodal tDCS applied over primary motor cortex (M1) - Dose: 1mA, 20 minutes + ( concomitantly) protocol of specific exercises for balance
  Interventions: Device: Transcranial direct current stimulation (tDCS); Other: Balance exercises
- Sham tDCS + Exercise (Sham Comparator): Sham tDCS applied over primary motor cortex (M1) - Dose: 1mA, 30 seconds ON, + (concomitantly) protocol of specific exercises for balance
  Interventions: Device: Transcranial direct current stimulation (tDCS); Other: Balance exercises

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — Transcranial direct current stimulation is a noninvasive technique of neuronal modulation.
Other: Balance exercises — Specific balance exercises, focused on balance, postural control and control of the center of gravity within the support base.

SUMMARY:
Neural control of posture depends on interaction of sensory and motor information from multiple structures, including the primary motor cortex (M1). Transcranial direct current stimulation (TDCS) improves postural control in children and adults with and without neurological disorders, however, additive effects to physical therapy treatment are still unknown, specifically balance exercises for children with balance deficit. The aim of this study is to identify the effects of adding anodic TDCS over M1 to exercises on postural control of children with balance deficit. This is a randomized, double-blind, controlled clinical trial.

DETAILED DESCRIPTION:
Maintaining body position and orientation is a complex and multifactorial task. Balance is defined as the ability to control and maintain the center of gravity or center of mass over the area of the support base. Postural control system aims (1) to maintain balance and postural orientation (2) to perform voluntary movement in static or dynamic circumstances and (3) to react to internal and external disturbances. Neural control of posture will be efficient when there is an interaction of sensory and motor information from multiple structures, and it will vary according to the age of the individuals, maturation of the structures involved, motor repertoire, neuromuscular synergies and musculoskeletal components, among others. The primary motor cortex (M1) has been persistently studied due to its complexity, numerous connections and direct involvement with motor control. Studies suggest that the main neural activity of M1 is to command muscle activity and optimize the effector system´s operation, producing a more uniform, efficient and coordinated motor response, including postural responses to mechanical disturbances.

When one of the organs involved in this function is compromised, regardless of the age of the individuals, whether due to injury or a change in functioning or integration, body oscillations happen. Historically, balance deficit (and consequent falls) are considered normal and acceptable in childhood, however, it is necessary to be careful with falls and their consequences in children with mobility or behavioral diseases. Physical therapy is essential in the rehabilitation of children and adults with balance deficit, with or without injury in nervous system. Currently, there is an increasing number of studies that have pointed Transcranial direct current stimulation (TDCS) as an efficient and safe device to modulate motor performance. To our knowledge, despite this growing number of studies, little is known about how much TDCS could add to an balance exercise protocol for children without structural damage in nervous system with balance deficit. Therefore, it is relevant to carry out studies in order to investigate and possibly elucidate the effects of TDCS on postural control and balance in children. Thus, the aim of this study is to identify the effects of adding anodic TDCS over M1 to exercises on postural control of children with balance deficit. This is a randomized, double-blind, controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* children of both sex
* aged between 6 -11 years old;
* assent of the child by the Term of Assent and acceptance of parents and / or guardians to participate in the study by signing the Free and Informed Consent Form;
* children with percentile <=5 in the MABC-2(Movement Assessment Battery for Children second edition) Motor Evaluation Battery and in the balance domain and <=25 in total score
* children with percentile <=9 in the MABC-2 Motor Evaluation Battery and in the balance domain and <=5 in total score

Exclusion Criteria:

* visual or auditory deficiencies; cardiopathies; rheumatic or orthopedic dysfunctions; neurological or psychiatric problems (except Attention Deficit Hyperactivity Disorder and Developmental Coordination Disorder).

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2020-06-20 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Displacement of COP (center of pressure) | through study completion, an average of 10 months
  AP (anteroposterior) displacement (cm), ML (mediolateral) displacement (cm), area of the displacement (cm2) and velocity of the displacement (cm/sec)

SECONDARY OUTCOMES:
Motor performance in dynamics balance tasks | through study completion, an average of 10 months
  TUG Test
Motor performance in balance scale (dynamic and static balance tasks) | through study completion, an average of 10 months
  Pediatric Balance Scale

CONTACTS AND LOCATIONS:
Overall Officials: Renata Hydee Hasue, Principal Investigator — Faculty of Medicine, University of São Paulo
Locations (1):
- Department of Physical Therapy, Communication Sciences and Disorders, and Occupational Therapy, Faculty of Medicine, University of São Paulo, São Paulo, Brazil